CLINICAL TRIAL: NCT03419689
Title: Biomarker Discovery Project in High Grade Serous Ovarian Cancer
Brief Title: Study Looking at Biomarkers in Ovarian Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BioDIVA (17-5467)
Record Dates: First submitted 2017-08-08; First posted 2018-02-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sample Collection (Experimental): The following samples may be collected during the study:
  * Tumour tissue samples
  * Blood samples
  * Ascites samples
  * Other fluids requiring drainage
  Interventions: Procedure: Tumour tissue collection; Procedure: Blood sample collection; Procedure: Ascites Collection; Procedure: Fluid Collection

INTERVENTIONS:
Procedure: Tumour tissue collection — Tumour tissue will be taken from samples already removed from surgery or biopsy or by new tumour biopsies:
  * At the time of diagnosis or progression
  * Any surgical procedures for management of tumour related medical conditions
  * At each subsequent relapse or disease progression
Procedure: Blood sample collection — Blood samples will be taken:
  * At the time of first diagnosis
  * About 1 week after starting any treatment
  * At each radiological response assessment
  * At each subsequent relapse or disease progression
Procedure: Ascites Collection — Ascites will be collected if paracentesis is required during any of the following time points:
  * At the time of diagnosis or progression
  * Any surgical procedures for management of tumour related medical conditions
  * At each subsequent relapse or disease progression
Procedure: Fluid Collection — Additional fluid will be collected at any time a procedure for clinical management that involves the drainage of fluid (i.e. thoracentesis, or drainage of cystic lesion) is required.

SUMMARY:
This is a sample study that will collect biological samples (blood, tumor tissue, ascites, and/or other fluids) from gynecological cancer patients for biomarker research. In addition, the results of the testing done on the samples will be given to the participant's treating physician who may use the information to guide treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of stage III or IV high grade serous ovarian, tubal or primary peritoneal cancer.
* Must be 18 years of age or older.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
* Have a life expectancy greater than or equal to 6 months.
* Able to provide adequate informed consent.
* Willing to undergo blood or fluid collection and tumour biopsy
* Patients enrolled at the time of surgery must agree to have part of their tumour used for the purpose of the study.
* Archival tissue must be available for patients that are enrolled at the time of progression.

Exclusion Criteria:

* Must not have early stage (I and II) high grade serous, tubal or primary peritoneal cancer.
* Must not have other tumour histology other than high grade serous.
* Must not have contraindication to tumour biopsy and/or blood sampling.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2028-06-08 (Estimated); Study Completion 2028-06-08 (Estimated)

PRIMARY OUTCOMES:
Genomic and immune signatures in terms of progression free survival | 10 years
  Short term (1-2 years) versus long term (5-10 years) survival
Genomic and immune signatures in terms of overall survival | 10 years
  Short term (1-2 years) versus long term (5-10 years) survival
Genomic and immune signatures in terms of response to treatments | 10 years
Genomic and immune signatures in terms of resistance to treatments | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (7):
- Canada (7):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario